CLINICAL TRIAL: NCT01450410
Title: Efecto Del ácido nicotínico Sobre la composición de Las lipoproteínas de Alta Densidad (HDL) y la función Del Endotelio Arterial en Los Pacientes Con cardiopatía isquémica Prematura y Concentraciones Elevadas de Colesterol-HDL
Brief Title: Nicotinic Acid Composition of HDL and Arterial Endothelium Function in Premature Coronary Heart Disease and High HDL
Acronym: 11MSP011
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated (halted prematurely) as recomended by the drug supplier and medical agencies
Sponsor: Xavier Pinto Sala (Other)
Responsible Party: Sponsor-Investigator, Xavier Pinto Sala, Principal Investigator, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: CompHDL2011
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2011-11

CONDITIONS: Dyslipidemias
Keywords: Dyslipemia, HDL composition
MeSH Terms: conditions — Dyslipidemias | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotinic Acid (Active Comparator)
  Interventions: Drug: Nicotinic acid
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotinic acid — Nicotinic acid / laropiprant (Tredaptive 1000 mg/20 mg modified-release tablets). Patients treated with nicotinic acid 1g/day receive one dose of one month and 2 g / day thereafter. Nicotinic acid treatment will last for 12 weeks.
  Other Names: Tredaptive
  Arms: Nicotinic Acid
Drug: Placebo — Placebo treatment will last for 12 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
Patients with premature ischemic heart disease (PIHD) and elevated levels of HDL-C present an altered composition of high-density lipoproteins (HDL) which is associated with a loss of their anti-atherogenic effects and of their arterial endothelium function.

Objectives: To analyse if the treatment with nicotinic acid (NA)/Laropiprant can correct the alterations of the HDL composition and endothelial function in patients with PIHD and elevated HDL-C.

Methods: A total of 46 subjects with PIHD who are stable in the 3 months prior to the Study, who continue in treatment with statins and have elevated concentrations of HDL-C (HDL-C ≥2.0mmol/L in females and ≥1.8mmol/L in males) and an LDL-C <100mg/dL. This is a double-blind, randomised Study; after 6 weeks of lifestyle stabilisation, the subjects will be treated with NA or placebo for 16 weeks. At the start and end of treatment, HDL composition will be studied through density gradient preparative ultracentrifuge separation and FBLC (fast protein liquid chromatography) and through the changes in vasodilation induced by the endothelium through ultrasound. Primary endpoint: change in the apoA1 content associated to treatment. Secondary endpoints: variations in the change of the brachial artery diameter with reactive hyperaemia and changes in the content of other lipid and protein components of HDL including apoA2, paraoxonase, amyloid A and LCAT. The changes in HDL composition and endothelial function will be assessed with an analysis of variance with repeated measurements and a 2x2 design.

ELIGIBILITY:
Inclusion Criteria:

* Being male or female
* Age > 25 years
* Have an episode of ischemic heart disease before 55 years in men and in women 65 years
* Serum HDL-C above the 90th percentile of the Spanish population: >=2.0mmol/L in women and >=1.8mmol/L in men (Gomez-Gerique JA, et al. Med Clin (Barc.). 1999, 113: 730-735.)
* Stable treatment with any statin in the past 6 weeks: simvastatin, atorvastatin, rosuvastatin, pravastatin or lovastatin.

Exclusion Criteria:

* Uncontrolled hypercholesterolemia or hypertriglyceridemia, LDL-C >2.6mmol/L or triglycerides >2.24mmol/L
* Patients with an episode of ischemic heart disease in the last 3 months
* Patients suffering from acute or chronic inflammatory diseases in the last 3 months
* Treatment with fibrates or omega-3 fatty acids.
* Treatment with steroids or immunosuppressive drugs
* Patients with a contraindication to Tredaptive (Hypersensitivity to the active substances or any of the excipients, significant or unexplained hepatic dysfunction, active peptic ulcer, arterial bleeding).
* Patients treated with drugs that may interact with Tredaptive (Midazolam).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Apo A1 of HDL | Baseline; 12 weeks
  The amount of Apo A1 as a marker of HDL composition.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Pintó, PhD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Unitat Funcional de Risc Vascular. Servei Medicina Interna. Hospital Universitari de Bellvitge., L'Hospitalet de Llobregat, Barcelona, Spain